CLINICAL TRIAL: NCT06501430
Title: Effects of Autogenic Inhibition and Reciprocal Inhibition on Pain, Range of Motion, Function and Sports Performance in Amateur Football Players With Shin Splints.
Brief Title: Effects of Autogenic Inhibition and Reciprocal Inhibition in Amateur Football Players With Shin Splints.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0484
Record Dates: First submitted 2024-07-09; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Shin Splint
Keywords: Football Players; Shin Splints; Pain; Sports performance
MeSH Terms: conditions — Medial Tibial Stress Syndrome; Pain

STUDY DESIGN:
Intervention Model Description: After recruitment and signing the informed consent, baseline readings of all study variables will be taken and all subjects will be assigned into 2 groups, GROUP A (received autogenic inhibition with conventional treatment) and GROUP B (received reciprocal inhibition with conventional physiotherapy treatment) randomly divided by computer-generated software.
Who Masked: Participant, Investigator
Masking Description: Subjects of both groups (Group A and B) will be kept unaware of the treatment type given to other group. All the information will be kept in lock and key, and will be accessible to author only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autogenic Inhibition (Experimental): Group 1 will receive Autogenic inhibition with conventional treatment. Autogenic inhibition will be applied to the muscles of the anterior tibial compartment, including Tibialis anterior, extensor hallucis longus, extensor digitorum longus (Perform Dorsi-Flexion), Lateral Tibial Muscles (Peronei), and posterior tibial muscles including, gastrocnemius, soleus and plantaris (Perform Plantarflexion).
  Interventions: Other: Heating Therapy; Other: Manual Soft tissue Release
- Reciprocal Relaxation (Experimental): Group 2 will receive reciprocal inhibition with conventional treatment. Reciprocal inhibition will be applied to the muscles of the anterior tibial compartment, including Tibialis anterior, extensor hallucis longus, extensor digitorum longus (Perform Dorsi-Flexion), Lateral Tibial Muscles (Peronei), and posterior tibial muscles including, gastrocnemius, soleus and plantaris (Perform Plantarflexion).
  Interventions: Other: Heating Therapy; Other: Manual Soft tissue Release

INTERVENTIONS:
Other: Heating Therapy — Heating Therapy will be performed on subjects along with PNF Exercises.
Other: Manual Soft tissue Release — Manual Soft tissue Release will be performed on subjects along with PNF Exercises.

SUMMARY:
This randomized controlled trial aims to compare the effectiveness of Autogenic Inhibition and Reciprocal Inhibition in treating shin splints among amateur footballers aged 18-30 from SA Gardens Football Club, Lahore. Participants will be recruited through non-probability convenient sampling and randomly assigned into two groups using random number sampling. A single-blind approach will be employed, with one group receiving Autogenic Inhibition treatment and the other receiving Reciprocal Inhibition treatment over a period of four weeks, with three sessions per week. The study will measure outcomes including pain alleviation, improvement in range of motion (ROM), enhanced function, and improved sports performance. This research seeks to provide insights into the benefits of muscle energy techniques for athletes with shin splints, contributing valuable knowledge to sports medicine and rehabilitation practices.

DETAILED DESCRIPTION:
Recent literature provides substantial evidence supporting the efficacy of muscle energy techniques (METs), including Autogenic Inhibition, for various musculoskeletal conditions across different populations. Robert F. et al. (2023) conducted a quasi-experimental study using a pre- and post-test design to compare Kalternborn grade III mobilization and METs in 30 patients, finding significant improvements in pain and neck function. Siddiqui M. et al. (2022) demonstrated in a randomized control trial that Autogenic Inhibition was more effective than Reciprocal Inhibition in improving pain, range of motion, and functional disability in patients with mechanical neck pain. Similarly, Osama M. et al. (2022) found Autogenic Inhibition to be the most effective among static stretching, AI-MET, and RI-MET for enhancing isometric muscle strength in neck pain patients. Majeed A. et al. (2021) showed that Autogenic Inhibition had better outcomes than static stretching for hamstring flexibility. Khaled H. Yousef et al. revealed that adding METs to conventional therapy significantly improved pain, impairment, and hip range of motion in patients with chronic discogenic sciatica. A systemic review by Thomas E. et al. (2019) confirmed METs' effectiveness in reducing chronic and acute pain and improving range of motion. Despite these positive findings, there is limited research on METs for sports-related conditions like shin splints. This study aims to fill this gap by examining the specific benefits and drawbacks of a structured MET program for shin splints in a sports environment, providing valuable insights for athletes in managing and preventing overuse and bone stress injuries efficiently.

ELIGIBILITY:
Inclusion Criteria:

1. Both genders.
2. Age 18-30 years.
3. Those who are actively taking part in sports from last 1 year.
4. Subjects who have NPRS scores from moderate pain (NPRS 4-6) to severe pain (NPRS 7- 10).
5. Subjects diagnosed with category 2 Shin splints through Shin splint scoring system (Male 2- 14, Female 6-16) and category 3 (Male 14-29, Female 17-29).

Exclusion Criteria:

1. History of Central or peripheral vascular disease.
2. History of lower limb fracture / Trauma (Any side) in last 6 months.
3. History of lower limb Surgery (Any side) in last 6 months.
4. History of any malignancy.
5. Leg length discrepancy.
6. Biomechanical imbalances.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-12-23 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Pain: Numeric Pain Rating Scale (NPRS) | 1st day and 12th week.
  NPRS is a reliable tool when measuring pain.
Ranges of Motion: Goniometery | 1st day and 12th week.
  The testing position will supine laying with foot in a resting position and towel rolled under ankle, the goniometer center will be on either of the malleolus. The proximal arm will be placed parallel to the ground or tibia/fibula. The distal arm will be moved with the movement of foot into dorsiflexion or plantarflexion.
Function: Lower Extremity Functioning Scale (LEFS) | 1st day and 12th week.
  LFS is reliable tool to measure lower extremity functional status. It will take 2-5 minutes with each subject to take th readings.
Performance: 60m yard test | 1st day and 12th week.
  1.60m yard test Athlete to sprint as fast as possible over 60 metres after warming up for 10 minutes. The assistant marks out a 60-metre straight section on the track with cones. The assistant gives the command "GO" and starts the stopwatch. The athlete sprints as fast as possible over the 60 metres. The assistant stops the stopwatch as the athlete's torso crosses the finishing line and records the time.
Performance: Yoyo Test | 1st day and 12th week.
  Yoyo test: Subject performs an appropriate warm-up. Use cones to mark out two lines 20 meters apart as per the diagram. The participants start with their foot behind one of the lines, and begin running when instructed. They continue running between the two lines, turning when signaled by the recorded beeps. After each minute or so, the pace gets quicker. If the line is not reached in time the subject must run to the line, turn and try to catch up with the pace within 2 more 'beeps. The test is stopped if the subject fails to catch up with the pace within the two ends.

CONTACTS AND LOCATIONS:
Overall Officials: Zohaib Imran, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Sports Board, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eime RM, Young JA, Harvey JT, Charity MJ, Payne WR. A systematic review of the psychological and social benefits of participation in sport for children and adolescents: informing development of a conceptual model of health through sport. Int J Behav Nutr Phys Act. 2013 Aug 15;10:98. doi: 10.1186/1479-5868-10-98. PMID 23945179
- [Background] Christakou A, Lavallee D. Rehabilitation from sports injuries: from theory to practice. Perspect Public Health. 2009 May;129(3):120-6. doi: 10.1177/1466424008094802. PMID 19514635
- [Background] Prieto-Gonzalez P, Martinez-Castillo JL, Fernandez-Galvan LM, Casado A, Soporki S, Sanchez-Infante J. Epidemiology of Sports-Related Injuries and Associated Risk Factors in Adolescent Athletes: An Injury Surveillance. Int J Environ Res Public Health. 2021 May 2;18(9):4857. doi: 10.3390/ijerph18094857. PMID 34063226
- [Background] Deshmukh NS, Phansopkar P. Medial Tibial Stress Syndrome: A Review Article. Cureus. 2022 Jul 7;14(7):e26641. doi: 10.7759/cureus.26641. eCollection 2022 Jul. PMID 35949792
- [Background] 5. Patel PY, Patil N. Prevalence of shin splint in recreational marathon runner. International Journal of Physiotherapy. 2020:37-41.
- [Background] Hanlon C, Krzak JJ, Prodoehl J, Hall KD. Effect of Injury Prevention Programs on Lower Extremity Performance in Youth Athletes: A Systematic Review. Sports Health. 2020 Jan/Feb;12(1):12-22. doi: 10.1177/1941738119861117. Epub 2019 Aug 7. PMID 31390306
- [Background] Newsham KR, Beekley MD, Lauber CA. A neuromuscular intervention for exercise-related medial leg pain. J Sport Rehabil. 2012 Feb;21(1):54-62. doi: 10.1123/jsr.21.1.54. Epub 2011 Nov 15. PMID 22104168
- [Background] Lee JH, Park SJ, Na SS. The effect of proprioceptive neuromuscular facilitation therapy on pain and function. J Phys Ther Sci. 2013 Jun;25(6):713-6. doi: 10.1589/jpts.25.713. Epub 2013 Jul 23. PMID 24259836
- [Background] Amako M, Oda T, Masuoka K, Yokoi H, Campisi P. Effect of static stretching on prevention of injuries for military recruits. Mil Med. 2003 Jun;168(6):442-6. PMID 12834132
- [Background] 10. Kumar P, Moitra M. Efficacy of muscle energy technique and pnf stretching compared to conventional physiotherapy in program of hamstring flexibility in chronic nonspecific low back pain. Indian J Physiother Occup Ther Int J. 2015;9(3):103.
- [Background] 11. Robert F, Anandh V, Arunachalam R, Kannan D, Kohilavani S, Thenmozhi M. A Comparative Study Between Kalternborn Grade Iii Mobilization And Muscle Energy Technique To Increase Range And Functional Ability Among Patients With Mechanical Neck Pain. Journal of Pharmaceutical Negative Results. 2023:3307-9.
- [Background] Siddiqui M, Akhter S, Baig AAM. Effects of autogenic and reciprocal inhibition techniques with conventional therapy in mechanical neck pain - a randomized control trial. BMC Musculoskelet Disord. 2022 Jul 25;23(1):704. doi: 10.1186/s12891-022-05668-0. PMID 35879756
- [Background] Osama M. Effects of autogenic and reciprocal inhibition muscle energy techniques on isometric muscle strength in neck pain: A randomized controlled trial. J Back Musculoskelet Rehabil. 2021;34(4):555-564. doi: 10.3233/BMR-200002. PMID 33523036
- [Background] 14. Majeed A, Mansoor SR, Arif AB, Yasin MM, Wasim M, Naeem F. Comparison of static stretching and muscle energy techniques on hamstring tightness in asymptomatic females. Foundation University Journal of Rehabilitation Sciences. 2021;1(1):19-23.
- [Background] 15. Yousef KH, Khalefa BM, Badawy MS, Foad A, Abdelmonem AMEG, Al-azab IMA-a. EFFECT OF MUSCLE ENERGY TECHNIQUES ON FUNCTIONAL ABILITIES IN PATIENTS WITH DISCOGENIC UNILATERAL SCIATICA. Turkish Journal of Physiotherapy and Rehabilitation.32:3.
- [Background] Thomas E, Cavallaro AR, Mani D, Bianco A, Palma A. The efficacy of muscle energy techniques in symptomatic and asymptomatic subjects: a systematic review. Chiropr Man Therap. 2019 Aug 27;27:35. doi: 10.1186/s12998-019-0258-7. eCollection 2019. PMID 31462989
- [Background] 17. White D. Muscle Energy Techniques as Part of a Comprehensive Plan of Care for a Patient with Hip and Knee Osteoarthritis: A Case Report. 2019.
- [Background] 19. Payla M, Gill M, Singal SK, Shah N. A Comparison of the Immediate and Lasting Effects between Passive Stretch and Muscle Energy Technique on Hamstring Muscle Extensibility. Indian Journal of Physiotherapy & Occupational Therapy. 2018;12(1).
- [Background] 20. Joshi R, Rathi M, Khandare S, Palekar TJ. Effect of muscle energy technique on pain and function in patients with sacroiliac dysfunction-experimental study. Int J Sci Res Educ. 2017;5(6):25-30.
- [Background] 21. Addala D, Kumar KS, Madhavi K. Effectiveness of Muscle Energy Technique on Pain and Range of Motion on Osteoarthrosis of Knee. Indian Journal of Physiotherapy and Occupational Therapy. 2013;7(4):29.
- [Background] Nussbaum ED, Gatt CJ Jr, Epstein R, Bechler JR, Swan KG, Tyler D, Bjornaraa J. Validation of the Shin Pain Scoring System: A Novel Approach for Determining Tibial Bone Stress Injuries. Orthop J Sports Med. 2019 Oct 30;7(10):2325967119877803. doi: 10.1177/2325967119877803. eCollection 2019 Oct. PMID 31696132
- [Background] de Bruijn JA, Wijns KCA, van Kuijk SMJ, Hoogeveen AR, Teijink JAW, Scheltinga MRM. Chronic exertional compartment syndrome in the differential diagnosis of peripheral artery disease in older patients with exercise-induced lower limb pain. J Vasc Surg. 2021 Jun;73(6):2114-2121. doi: 10.1016/j.jvs.2020.11.027. Epub 2020 Dec 2. PMID 33278541
- [Background] Ferraz MB, Quaresma MR, Aquino LR, Atra E, Tugwell P, Goldsmith CH. Reliability of pain scales in the assessment of literate and illiterate patients with rheumatoid arthritis. J Rheumatol. 1990 Aug;17(8):1022-4. PMID 2213777
- [Background] 26. Magee D. Orthopaedic physical assessment WB Saunders. pg. 2002;478:483-631.
- [Background] Binkley JM, Stratford PW, Lott SA, Riddle DL. The Lower Extremity Functional Scale (LEFS): scale development, measurement properties, and clinical application. North American Orthopaedic Rehabilitation Research Network. Phys Ther. 1999 Apr;79(4):371-83. PMID 10201543
- [Background] Altmann S, Ringhof S, Neumann R, Woll A, Rumpf MC. Validity and reliability of speed tests used in soccer: A systematic review. PLoS One. 2019 Aug 14;14(8):e0220982. doi: 10.1371/journal.pone.0220982. eCollection 2019. PMID 31412057
- [Background] Grgic J, Oppici L, Mikulic P, Bangsbo J, Krustrup P, Pedisic Z. Test-Retest Reliability of the Yo-Yo Test: A Systematic Review. Sports Med. 2019 Oct;49(10):1547-1557. doi: 10.1007/s40279-019-01143-4. PMID 31270753